CLINICAL TRIAL: NCT07060482
Title: Diagnostic Performance of Combined Assays for Gastrin-17, Pepsinogen and Anti-helicobacter Pylori Antibodies for Diagnosing Gastric Atrophy.
Brief Title: Gastrin, Anti-helicobacter Pylori and Pepsinogen Diagnostic Accuracy Study
Acronym: GAP-DA
Status: Not yet recruiting | Type: Observational
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Principal Investigator, Eoghan Burke, Specialist Registrar in Oesophagogastric Surgery, Royal College of Surgeons, Ireland
Other Study IDs: 24-248
Record Dates: First submitted 2025-03-21; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Gastric Atrophy
Keywords: gastric atrophy; pepsinogen; gastrin 17; anti-helicobacter pylori antibodies; gastroscopy
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients presenting for routine diagnostic gastroscopy.: Patients presenting for routine diagnostic gastroscopy.
  Interventions: Diagnostic Test: Panel of biomarkers including Gastrin 17, pepsinogen 1 and 2, and anti-helicobacter pylori antibodies.

INTERVENTIONS:
Diagnostic Test: Panel of biomarkers including Gastrin 17, pepsinogen 1 and 2, and anti-helicobacter pylori antibodies. — This study will be assessing the diagnostic accuracy of this panel of biomarkers for diagnosing gastric atrophy in the Irish population for the first time. This reflects the assessment of these biomarkers in diagnosing gastric atrophy in a low-risk Western population.

SUMMARY:
This research study is taking place to find out if a simple blood test can diagnose inflammation in the stomach. Prolonged inflammation in the stomach can lead to Ulcers and even Cancer in the long run.

Currently, a camera test is needed to identify inflammation in the stomach. The method being tested in this study may be able to do this using just a pinprick of blood.

If this test proves to be good at diagnosing inflammation in the stomach with just a pinprick of blood, it may be used in the future to decide who actually needs to have a full camera test done or not. This could really improve the waiting lists for these camera tests in the future. It may also mean that we can identify problems at an earlier stage.

DETAILED DESCRIPTION:
Gastric atrophy (GA), also referred to as atrophic gastritis, is a pre-neoplastic lesion in the development of intestinal-type gastric cancer (GC). It is defined as the loss of the normal glandular architecture of the stomach. It forms part of the so-called "Correa cascade", first described in 1988. This cascade posits that intestinal-type GC develops along a defined pathway of pre-neoplastic lesions. The initiation of this pathway is triggered by chronic inflammation affecting the gastric mucosa. The cause of this chronic inflammation is most commonly Helicobacter Pylori, although chronic autoimmune gastritis accounts for a minority of cases. The chronic inflammation over time causes the loss of the normal glandular architecture characteristic of gastric atrophy. With the ongoing presence of the initiating factor and persistence of the chronic inflammatory phenotype, the GA can progress to intestinal-type metaplasia and then to dysplasia and, ultimately, intestinal-type gastric cancer.

The precise risk of progression to GC in those with GA is poorly understood, particularly in lower-risk Western countries such as Ireland. In higher-risk countries such as Japan and South Korea, the reported risk may be as high as 0.1 to 0.3% per year. This is similar to the rates of malignant progression seen in low-risk colorectal adenomas and the risk seen in non-dysplastic Barrett's. This has prompted increased interest in the concept of surveilling patients with GA in the hopes of earlier identification of GC. Indeed, there is evidence to suggest that if Helicobacter Pylori is eradicated in patients with GA, the Correa cascade can be halted, and the risk of developing GC can be greatly reduced.

The British Society of Gastroenterology addressed this issue in their guideline document published in 2019. The guideline addresses several issues concerning managing patients at risk of developing Gastric Adenocarcinoma. Central to this is the concept of managing patients with GA. The guideline advocates for increased endoscopist awareness of the macroscopic features of the atrophic stomach. When recognised, the endoscopist should then take targeted biopsies as per the Updated Sydney System. This biopsy regimen involves taking Biopsies from the antrum, both lesser and greater curvature, the incisura and the gastric body again, both lesser and greater curvature. These biopsies should be sent to the lab in separately labelled specimen jars. The histological assessment should then be conducted using the Operative link for Gastritis assessment system, also known as the OLGA system. This classifies the severity of GA into 4 subtypes. There is evidence to suggest that patients with OLGA stage 3 or 4 GA should enter a 3-yearly surveillance program. This pathway is well established and in practice.

The issue currently, however, remains identifying patients with GA. With ever-increasing waiting lists for endoscopic procedures and growing numbers of dyspeptic patients, there is a need to triage referrals to increase the diagnostic yield from oesophagogastroduodenoscopies (OGDs). The use of Biomarkers to identify patients at risk of GA is one such potential pathway.

A panel of biomarkers (commercially available as the GastroPanel), including pepsinogen 1, pepsinogen 2, Gastrin 17, and IgG antibodies to Helicobacter pylori, has been shown to predict GA in high-risk regions. However, their efficacy in identifying GA in lower-risk Western cohorts of patients is less well known. This combination of biomarkers is instructive of the morphological state of the gastric mucosa. Pepsinogen 1 is produced predominantly by the chief cells of the oxyntic mucosa of the corpus and fundus of the stomach. Pepsinogen 2 is similarly produced by the chief cells but also by neck mucous cells, which are found in the oxyntic mucosa and the pyloric mucosa of the antrum and pyloric canal. Thus, in the setting of GA of the oxyntic mucosa, pepsinogen 1 levels will decrease to a greater extent than pepsinogen 2 levels. Gastrin 17 is a peptide produced by the G cells of the diffuse neuroendocrine system located in the pyloric mucosa of the antrum and pyloric canal. Decreased levels of Gastrin 17 are seen in the setting of GA of the pylorus. Thus, by evaluating the levels of these biomarkers, it may be possible to predict both the presence and topological extent of GA.

An assessment of these biomarker levels, in concert with the patient's clinical history, including symptoms and risk factors, could then be used to triage OGD waiting lists. Patients with biomarker levels suggestive of GA may then be prioritised for an OGD.

Previous testing algorithms for these biomarkers involved the drawing of a serum sample and then assessment of the biomarker levels via an enzyme-linked immunosorbent assay (ELISA) test. This may have limited application in the clinical setting, given the lab space and experience needed to conduct this test. However, recent improvements in point-of-care testing technology, including the development of an immunological lateral flow testing method for these biomarkers (GastroPanel QuickTest), raise the possibility of a useable clinic-based test. The most recent iteration of this device is based on the acquisition of a pinprick of whole blood from the patient's finger. This is similar in practice to the testing method of blood sugar levels, which is routinely done prior to various tests, including OGDs.

We intend to assess the diagnostic accuracy of this test against the gold standard of endoscopically obtained gastric mucosa biopsies in patients presenting for OGDs in Beaumont Hospital, Dublin, Ireland. Patients will be prospectively identified and invited to participate in the study following informed consent. When they arrive for their OGD, a pinprick of whole blood will be obtained prior to their OGD. The immunological lateral flow testing machine is portable and will be in the Endoscopy room. The test will be run while the patient has their OGD as planned. Routine biopsies from the oxyntic and pyloric mucosa will be obtained. The lateral flow test results will then be compared to the histological results of the biopsies to assess the diagnostic accuracy of both the biomarkers and the lateral flow testing method.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for a routine diagnostic gastroscopy.

Exclusion Criteria:

* Patients presenting for a therapeutic procedure such as dilations or stenting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to evaluate our primary objective of determining the diagnostic accuracy of the point of care immunological lateral flow test in diagnosing Gastric atrophy, we will recruit 240 patients who are presenting to the endoscopy day unit for diagnostic gastroscopy in Beaumont Hospital, Dublin.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Diagnosed with Gastric Atrophy by GastroPanel QuickTest Compared to Histology | This diagnostic accuracy assessment will occur simulatneously at the time of the patients gastroscopy with both the blood sample and gastric biopsies being taken at that time.
  Diagnostic accuracy of the GastroPanel QuickTest (Biohit) for detecting gastric atrophy, assessed by comparing the combined biomarker panel result-including Gastrin-17, Pepsinogen 1, Pepsinogen 2, and anti-Helicobacter pylori IgG antibodies-against the histological diagnosis of gastric atrophy from gastric biopsies. Accuracy metrics will include sensitivity, specificity, positive predictive value, and negative predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Eoghan Burke, MD, Principal Investigator — Royal college of Surgeons in Ireland

IPD SHARING:
Plan to Share IPD: Undecided